CLINICAL TRIAL: NCT00636584
Title: Does Sodium Nitroprusside Infusion Affect Thyroidal Function in Patients Undergoing Coronary Artery Bypass Grafting, a Prospective Randomized Clinical Trial.
Brief Title: Clinical Study Investigating the Effect of Sodium Nitroprusside Infusion on Thyroidal Function
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kavaklıdere Umut Hospital (Other)
Collaborators: Ankara University (Other)
Responsible Party: Kavaklıdere Umut Hastanesi, Kavaklıdere Umut Hospital, department of cardiovascular surgery
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2008-0048
Record Dates: First submitted 2008-03-07; First posted 2008-03-14 (Estimated); Last update posted 2008-03-14 (Estimated); Status verified 2008-03

CONDITIONS: Nitroprusside; Thyroid Hormones
Keywords: sodium nitroprusside; thyroid hormones; thoracic surgery
MeSH Terms: interventions — Nitroprusside

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): arm1: sodium nitroprusside group
  Interventions: Drug: sodium nitroprusside
- 2 (Placebo Comparator): arm2: control group,saline infused instead of sodium nitroprusside
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: sodium nitroprusside — sodium nitroprusside infusion at 1 microgram/kg/min dose during rewarming period of cardiac operations
  Other Names: nipruss
  Arms: 1
Drug: placebo — placebo
  Arms: 2

SUMMARY:
Whether use of SNP during cardiac surgery has any effect on thyroid function has not yet been investigated in humans. The aim of this study was to investigate the effects of SNP administration during the rewarming period of cardiac operations on circulating levels of thyroid hormones.

ELIGIBILITY:
Inclusion Criteria:

Patients without history of:

* thyroidal disease
* hypertension
* pulmonary disease
* peripheral vascular disease
* stroke
* recent myocardial infarction within the week prior to operation
* unstable angina pectoris
* liver or kidney dysfunction
* morbid obesity
* cachexia
* sulfonylurea intake

Exclusion Criteria:

* Patients who needed positive inotropic pharmacologic support during or after the operation
* Patients who developed atrial fibrillation in the post operative period requiring amiodarone therapy
* In addition, patients receiving any medication known to interfere with any step of thyroid hormone metabolism such as

  * amiodarone
  * propranolol
  * furosemide
  * non-steroidal anti-inflammatory agents
  * steroids
  * estrogens
  * antacids
  * diphenylhydantoin
  * spironolactone

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-02 (Actual); Study Completion 2008-03 (Estimated)

PRIMARY OUTCOMES:
free T3 | on admission, prior to operation, at the beginning of CPB, following CPB, at first, third and fifth postoperative days

SECONDARY OUTCOMES:
total T3 | on admission, prior to operation, at the beginning of CPB, following CPB, on the first, third and fifth postoperative days

CONTACTS AND LOCATIONS:
Overall Officials: alp aslan, md, Study Director — kavaklıdere Umut Hastanesi, Turkey
Locations (1):
- Kavaklıdere Umut Hastanesi, Ankara, Turkey (Türkiye)

REFERENCES:
- See also: home page of kavaklidere umut hospital — http://www.cityhospital.com.tr/